CLINICAL TRIAL: NCT02802228
Title: A Randomized, Double-blind, Placebo-controlled Pilot Study to Assess the Safety and Efficacy of Ifetroban for the Treatment of Portal Hypertension in Cirrhotic Patients
Brief Title: Study to Assess Safety and Efficacy of Ifetroban for Treatment of Portal Hypertension in Cirrhotic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPI-IFE-005
Record Dates: First submitted 2016-06-09; First posted 2016-06-16 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-01

CONDITIONS: Portal Hypertension; Liver Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis | interventions — ifetroban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ifetroban (Experimental): 90 day course of oral ifetroban following intravenous loading dose
  Interventions: Drug: Ifetroban
- Placebo (Placebo Comparator): 90 day course of placebo following intravenous dose of 5% dextrose in water (D5W)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ifetroban — thromboxane prostanoid receptor antagonist delivered as infusion and oral capsule
  Arms: Ifetroban
Drug: Placebo — matched placebo delivered as infusion and oral capsule
  Arms: Placebo

SUMMARY:
This placebo-controlled study will assess the safety and efficacy of a 90-day course of treatment with ifetroban for portal hypertension in cirrhotic patients

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis
* baseline hepatic venous pressure gradient (HVPG) >= 8 mmHg and <= 18 mmHg
* stable liver function enzymes

Exclusion Criteria:

* portal or splenic vein thrombosis
* Transjugular intrahepatic portosystemic shunt (TIPS) or portocaval shunt
* variceal bleed in last 2 months
* hemodialysis
* Child-Pugh Score >= 12
* Model for End-stage Liver Disease- Sodium score (MELD-Na) >= 20
* Acute kidney injury, Chronic kidney disease and/or Serum Creatinine >= 2.0 mg/dL
* current alcohol consumption > 2 drinks per day
* Platelet count (PLT) < 60 x 10^3/microliter (uL)
* A change in statin therapy in the last 3 months
* Current Hepatitis Virus B or C (HBV or HCV) therapy; or planned initiation of therapy during the treatment period
* Myocardial infarction within 30 days
* History of bleeding diathesis or current (within previous 14 days) or planned use of anticoagulant or antiplatelet drugs including aspirin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Rockey, MD, Principal Investigator — Medical University of South Carolina
Locations (6):
- United States (6):
  - Tampa General Medical Group, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ifetroban | Placebo
Started | 20 | 10
Completed | 15 | 10
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 90 day course of placebo following intravenous dose of D5W
  Placebo: matched placebo delivered as infusion and oral capsule
- Total: Total of all reporting groups
Arm/Group | Ifetroban | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (8.1) | 58.2 (9.1) | 55.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 18 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 10 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Primary Cirrhosis Etiology [Count of Participants; unit: Participants]
  Hepatitis B only | 0 | 0 | 0
  Hepatitis C only | 2 | 3 | 5
  Hepatitis B and C | 1 | 0 | 1
  Non-alcoholic Steatohepatitis | 8 | 3 | 11
  Alcoholic | 4 | 4 | 8
  Auto-immune | 3 | 0 | 3
  Cryptogenic | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety (Incidence and Severity of Adverse Events)
Description: Incidence is measured as the total number of adverse events reported during the treatment and follow-up period for each treatment group.
Time Frame: Through 97 days (90 days treatment and 7 days follow-up)
Measure: Number; unit: Number of adverse events
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 20 | 10
Number of adverse events | 23 | 2

2. Primary Outcome: Safety (Severity of Adverse Events)
Description: The severity of each event is reported by the investigator according to the following protocol/CTCAE definitions: Grade 1-Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2-Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living; Grade 3-Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4-Life-threatening consequences; urgent intervention indicated; Grade 5-Death related to adverse event.
Time Frame: Through 90 days treatment and 7 days follow-up
Measure: Count of Units; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 20 | 10
Number analyzed (Adverse Events) | 23 | 2
Adverse Events
  Grade 1 (mild) | 11 | 1
  Grade 2 (moderate) | 8 | 0
  Greade 3 (severe) | 4 | 1
  Grade 4 (life-threatening) | 0 | 0
  Grade 5 (death) | 0 | 0

3. Secondary Outcome: Change in Hepatic Venous Pressure Gradient (HVPG)
Description: The HVPG will be measured through Day 90 and will be compared to baseline
Time Frame: Baseline and 90 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 15 | 10
mmHg | 1.6 (3.7) | -0.1 (2.7)

4. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: AST values through Day 90 will be compared to baseline
Time Frame: Baseline and 90 days
Population: The analysis was performed on all subjects that had data available for the Baseline to Day 90 comparison.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 17 | 10
U/L | -1.2 (9.1) | 4.2 (12.9)

5. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: ALT values through Day 90 will be compared to baseline
Time Frame: Baseline and 90 days
Population: The analysis was performed on all subjects that had data available for the Baseline to Day 90 comparison.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 17 | 10
U/L | -4.8 (7.4) | 2.2 (9.1)

6. Secondary Outcome: Aspartate Aminotransferase/Platelet Ratio (APRI)
Description: The Aspartate Aminotransferase/Platelet Ratio through Day 90 will be compared to baseline
Time Frame: Baseline and 90 days
Population: The analysis was performed on all subjects that had data available for the Baseline to Day 90 comparison.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 16 | 10
ratio | 0.84 (0.52) | 0.98 (0.61)

7. Secondary Outcome: Variceal Bleeds (Occurrence of Variceal Bleeds)
Description: The number of variceal bleeds during the treatment and follow-up periods will be evaluated
Time Frame: Through Day 97
Measure: Number; unit: events of variceal bleeding
Arm/Group | Ifetroban | Placebo
Number analyzed (Participants) | 20 | 10
events of variceal bleeding | 0 | 1

ADVERSE EVENTS:
Time Frame: 90 days of investigational treatment and 7 days of follow-up
Arm/Group | Ifetroban | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/10
Other Adverse Events (participants affected / at risk) | 10/20 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ifetroban (N=20) | Placebo (N=10)
Ascites (Hepatobiliary disorders) | 1 (2) | 0 (0)
oesophageal varices haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ifetroban (N=20) | Placebo (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eccymosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Petechiae (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Dental discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Subacute cutaneous lupus erythematosus (Immune system disorders) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thromboelastogram (Investigations) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo positional (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT02802228/Prot_SAP_000.pdf